CLINICAL TRIAL: NCT05454982
Title: Effect of the Different Pressure Settings of a Continuous Cold-flow Cryocompression Device on Skin Temperature of the Knee: a Randomised Crossover Trial
Brief Title: Effect of Pressure on Skin Temperature When Using a Cryocompression Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Winchester (Other)
Collaborators: Physiolab Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HWB_REC_ 220530_Faulkner
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low pressure (Experimental): Participants will wear the cryocompression device for 30 minutes while ice-water at a temperature of 8℃ and a static pressure of 25 mmHg is applied to the lower limb by the cuff.
  Interventions: Device: Cryocompression
- Medium pressure (Experimental): Participants will wear the cryocompression device for 30 minutes while ice-water at a temperature of 8℃ and an intermittent pressure of 25-50 mmHg is applied to the lower limb by the cuff.
  Interventions: Device: Cryocompression
- High pressure (Experimental): Participants will wear the cryocompression device for 30 minutes while ice-water at a temperature of 8℃ and an intermittent pressure of 25-75 mmHg is applied to the lower limb by the cuff.
  Interventions: Device: Cryocompression

INTERVENTIONS:
Device: Cryocompression — A cryocompression device will be attached to the lower limb of participants using a cuff spanning from the mid-thigh to mid-calf. The device will circulate ice-water at a constant temperature of 8℃ throughout each test session. Depending on the condition, the cuff will also apply varying levels of pressure for the duration of each test. Each test session will last for 30 minutes. Participants will take part in all conditions, with at least 24 hours rest in between test sessions. Skin temperature around the knee will be measured prior to the cryocompression device being applied; every 5 minutes during the 30 minute test; and every 5 minutes after the test until skin temperature >15℃.

SUMMARY:
Cryotherapy after surgery is widely utilised and has numerous practical applications for post-operative rehabili-tation. Previous research has suggested that during cold therapy, the skin temperature of the knee should be reduced to 10-15°C to maximise the therapeutic benefits of cooling while avoiding the risk of cold injuries such as nerve damage and frostbite (Wilke and Weiner, 2003; Bleakley, McDonough and MacAuley, 2004). The degree to which the pressure applied by a cuff to the knee has an effect on the achieved skin temperature of the treatment area is unknown.

The aim of this study is to determine the effect that different pressure settings have on skin temperature around the knee during a 30-minute cryocompression treatment.

DETAILED DESCRIPTION:
This prospective randomised crossover trial will recruit healthy adult volunteers from a university population to participate. To avoid the involvement of individuals with unequal relationships, participants will be recruited through the form of advertisements on staff and student noticeboards, and through an email invitation sent to students within the faculty that the study will take place. A power analysis demonstrated that a total of 30 participants would be required to achieve a power of 0.8 and alpha error probability of 0.05 for a small-medium effect size of f=0.2. Each participant will take part in each condition within the study in order to eliminate the risk of demographic factors confounding the results: Conditions will be conducted in a random order and will be named: A, B, and C. These conditions will involve the device being worn while ice-water is circulated through the knee sleeve at a maintained temperature of 8°C with a pressure of either 25 mmHg, 25-50mmHg, or 25-75 mmHg, respectively. Randomisation will be performed using a computer random number generator. Each testing session will take 45-60 minutes to complete, with at least 24 hours between tests with the same participant. In total, participants will be giving around 3 hours across 3 days to complete their participation.. Participants will not be compensated for taking part in the study, nor will they be charged.

All eligible participants will first be required to provide informed consent prior to their participation in the study. Once this has been obtained, participants will each attend a single testing session that should last no longer than 60 minutes. The height and mass of the participants will first be measured in order to calculate BMI, and participants' age and sex will be recorded to allow for later analysis to determine any confounding influence of these factors on the results.

Participants will be required to remain in a seated position with their leg in full extension and elevated, parallel to the floor, for the duration of each test session. The leg that will be used for the study will be randomly selected for each participant, and will remain the same for each condition. Skin temperature will be measured using a thermocouple, which will be attached with tape 20 mm distal to the patella. The Physiolab S1 cryocompression device will then be attached to the leg of the participant and the test will begin. Depending on the condition to which a participant has been assigned for a given test, the S1 will maintain the temperature of the water flowing through the device while applying one of three different pressures.

The temperature of the skin will be measured using a k-type thermocouple attached to an infrared thermometer immediately prior to the application of the S1 device, and then every 5 minutes for the duration of the test. The cuff will be worn for 30 minutes as per the manufacturer guidelines for cold therapy treatments. After 30 minutes, the cuff will be removed. If the temperature of the skin has been reduced to within 10-15℃, skin temperature will continue to be monitored every 5 minutes after the cuff has been removed until it rises above 15℃, at which point the test will end. This will allow for the total time to be measured that skin temperature re-mains within the target therapeutic range as a result of a single application of the cryocompression device. If the skin temperature is not reduced to within 10-15℃ while the cuff is worn, then the test will end after the cuff is removed at 30 minutes. Upon completion of the test, the temperature sensor will be removed from the leg of the participant; thus completing their participation in the test. Once each participant has taken part in all conditions, they will have completed their participation in the study.

The data will be analysed to detect any differences during testing compared to baseline measures, and between groups. All data will be first subjected to a Kolmogorov-Smirnov test to assess whether they are normally distributed. A repeated measures analysis of variance will be performed on all normally distributed data. A Friedman test will be performed on any data that are not normally distributed.

There is a low risk of cold injury to participants if their skin temperature reduces to <10℃. Skin temperature will be monitored every 5 minutes throughout the study and testing will be terminated if a participant's skin temperature dips below this threshold. Therefore, the risk to participants in this study is minimal.

Participants have the right to withdraw themselves and any collected data from the study at any time during and after their participation, without having to give a reason. They also have the right to terminate a test session at any time. Testing shall also be terminated as a result of any adverse reactions that emerge. Adverse reactions (e.g. pain) to the testing protocol are not expected due to the low-risk nature of the study, however any that occur shall be recorded and monitored until things return to baseline/normal. In order to monitor any pain/discomfort that might occur, a Visual Analogue Scale (0-10 scale) will be within sight of the participant at all times during testing: a test will be terminated if reported pain/discomfort exceeds 5/10, though none is expected. Any reported pain (or other adverse reactions) shall be stored along with the data collected for that participant. If a test is terminated for a reason that could be mitigated in future, participants will be offered the opportunity to repeat the test another day, should they wish to continue taking part in the study. If a test is terminated due to an adverse reaction that can not be mitigated in future, the participant (and any collected data) will be thanked for their time and withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age.

Exclusion Criteria:

* BMI >40 kg/m2
* History of nerve damage or sensory deficit in the lower limbs (including frostbite)
* Hypersensitivity to cold, including hives
* Active inflammation or pain of the knee
* History of thrombosis, embolism, or other conditions related to impaired peripheral circulation
* Suffering from diagnosed diabetes, multiple sclerosis, rheumatoid arthritis, spinal cord injury, cardio-vascular disease, hypertension, Raynaud disease, cryoglobulinemia, or haemoglobinuria
* Confirmed or suspected tissue infection, an unstable fracture, a skin condition, or a tumour in the treatment area
* Cognitive impairment or communication barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Skin temperature | up to 14 days
  Skin temperature will be measured using a thermocouple positioned 20 mm distal to the patella. This sensor will be attached prior to the cryocompression device being applied, and will remain in place until the testing session is complete and skin temperature is >15℃. (The therapeutic skin temperature range for cryotherapy is thought to be 10-15℃). Temperature will be measured prior to the cryocompression device being applied; every 5 minutes during the test; and every 5 minutes after a test until the skin temperature reaches >15℃.

CONTACTS AND LOCATIONS:
Overall Officials: James Faulkner, PhD, Principal Investigator — University of Winchester
Locations (1):
- Physiology Laboratory, Winchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared outside of the researchers directly involved in the data collection itself.

REFERENCES:
- [Background] Wilke B, Weiner RD. Postoperative cryotherapy: risks versus benefits of continuous-flow cryotherapy units. Clin Podiatr Med Surg. 2003 Apr;20(2):307-22. doi: 10.1016/S0891-8422(03)00009-0. PMID 12776983
- [Background] Bleakley C, McDonough S, MacAuley D. The use of ice in the treatment of acute soft-tissue injury: a systematic review of randomized controlled trials. Am J Sports Med. 2004 Jan-Feb;32(1):251-61. doi: 10.1177/0363546503260757. PMID 14754753
- [Background] Fang L, Hung CH, Wu SL, Fang SH, Stocker J. The effects of cryotherapy in relieving postarthroscopy pain. J Clin Nurs. 2012 Mar;21(5-6):636-43. doi: 10.1111/j.1365-2702.2010.03531.x. Epub 2011 Feb 20. PMID 21332855
- [Background] Waterman B, Walker JJ, Swaims C, Shortt M, Todd MS, Machen SM, Owens BD. The efficacy of combined cryotherapy and compression compared with cryotherapy alone following anterior cruciate ligament reconstruction. J Knee Surg. 2012 May;25(2):155-60. doi: 10.1055/s-0031-1299650. PMID 22928433
- [Background] Selfe J, Hardaker N, Whittaker J and Hayes C. An investigation into the effect on skin surface temperature of three cryotherapy modalities. Thermology International. 2009; 19(4): 121-126.